CLINICAL TRIAL: NCT06415188
Title: The Effect of Therapeutic Play on Pre-Treatment Pain, Fear, Anxiety and Physiological Parameters and Parents' Satisfaction
Brief Title: The Effect of Therapeutic Play on Pain, Fear, Anxiety and Physiological Parameters and Parents' Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Sibel Küçükoğlu, Prof, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SelcukUni2544
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Child Behavior; Pain, Acute; Anxiety and Fear
Keywords: Pain; anxiety; children; nursing; therapeutic play
MeSH Terms: conditions — Child Behavior; Acute Pain; Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: This study was conducted on children aged 3-6 years. The study was completed with a total of 40 children and parent pairs in the experimental and control groups. Simple randomization method was used in the study. The randomization table for which group the children would be in was made by an independent statistician. Letters A and B were used to represent the experimental and control groups. Which letter represented which group was determined by lottery. While therapeutic play intervention was applied in the experimental group, routine intervention was applied in the control group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic play group (Experimental): Children in the experimental group received a therapeutic video game intervention in addition to the pre-treatment routine.
  Interventions: Behavioral: Video game with headset
- Control Group (No Intervention): Children in the control group underwent routine clinical practice. No other intervention was performed.

INTERVENTIONS:
Behavioral: Video game with headset — Half an hour before the first treatment in the morning, the screens around the patients' beds were closed by the researcher. The child was asked to choose one of the introduced games and the game he/she chose from the tablet was turned on. Children were asked to wear headphones for sound isolation and the sound was adjusted at the appropriate decibel setting. Half an hour before the treatment, children were allowed to play the video game until the treatment without any different warning. Physiologic Parameter Assessment Form, Child Anxiety and Fear Scale, Child Pain Scale were filled by the researcher 1 minute before and 1 minute after the procedure. Finally, Parental Satisfaction Scale was completed at the end of the intervention.
  Arms: Therapeutic play group

SUMMARY:
In this study, the effect of the therapeutic game applied before treatment on pain, fear, anxiety and physiological parameters and the satisfaction of the parents was investigated.

DETAILED DESCRIPTION:
Therapeutic play is defined as activities structured in accordance with children's age and development, or as a set of interventions to improve the well-being of children in the hospital environment. This method reduces the stress of illness or hospitalization, uses play as a means of self-expression and supports the development of positive coping mechanisms in pediatric patients. In the literature, it is seen that therapeutic play methods such as listening to music, drawing, reading stories, puppets, dolls, virtual reality tools, cartoon applications, watching videos and playing video games are used to reduce the child's pain and anxiety about invasive procedures. Studies conducted to reduce the interactions between children in the same environment during their treatment and care are quite limited. No study has been found to examine the effect of methods that jointly block/reduce vision and hearing during treatment and care on anxiety, fear and pain in children treated together in pediatric clinics.

ELIGIBILITY:
For the Child;

Inclusion Criteria:

* Being in the 3-6 age group,
* At least one day of inpatient treatment in the pediatric clinics of Selçuk Medical Faculty Hospital
* At least one invasive intervention in the treatment plan
* To be able to understand and speak Turkish
* Staying in a room with at least two beds

Exclusion Criteria:

* Having a neurological disorder
* Not having a parent as a companion
* Receiving oral treatment only
* Hearing and vision problems
* Single bed capacity room or isolated room

For the Parent

Inclusion Criteria:

* Staying with their child as a constant companion
* To be able to understand and speak Turkish
* Accepting to participate in the study

The exclusion criteria:

* Not staying with your child all the time

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Descriptive Characteristics Information Form | First measurement: 30 minute before treatment
  A descriptive characteristics information form for parents and children was prepared by the researchers in line with the literature and the data of both the experimental and control groups were collected before the intervention.
Physiological Parameter Monitoring Form | First measurement: 1 minute before treatment
  The descriptive characteristics form was based on a literature review by the investigator. Heart rate (min), oxygen saturation (SpO2%), blood pressure (mmHg) and respiratory rate (min) were measured 1 minute before treatment administration.
Children's State Anxiety and Children's Fear Scale | First measurement: 1 minute before treatment
  Children's State Anxiety and Children's Fear Scale was developed by McMurtry et al. in 2011. The scale was designed to measure the fear levels of children aged 4-10 years. The scale was translated into Turkish by Gerçeker et al. in 2018 and the validity-reliability coefficient was found to be 0.89. The scale score is formed by scoring five drawn facial expressions (0=no fear to 4=severe fear) shown visually to the child. Anxiety and fear scores of the child were scored one minute before the treatment.
Visual Analog Scale | First measurement: 1 minute before treatment
  Visual Analog Scale (VAS) was developed by Wong and Baker in 1988. Patients' pain levels are evaluated by scoring with facial expressions. It is used in children who have the ability to communicate and are conscious. The scale has 6 faces that are scored between 0 and 5. In scoring, the child chooses the face that best expresses him/her and "0" indicates no pain, "1" indicates a little pain, "2" indicates a little more pain, "3" indicates more pain, "4" indicates quite a lot of pain and "5" indicates the most severe pain level. One minute before the treatment, the child's pain is scored by VAS.
PedsQL Health Care Satisfaction Scale | First measurement: After treatment
  The PedsQL Health Care Satisfaction Scale was developed by J.W. Varni in 1999. Turkish adaptation of the scale was conducted by Ulus and Kublay in 2012. The scale consists of 25 items with 6 subheadings: emotional support, information, general satisfaction, communication, family involvement and technical skills. The scale is on a five-point scale and each item is rated on a scale of 0 to 4 and is evaluated as "Never satisfied (0)", "Sometimes satisfied (1)", "Most of the time satisfied (2)", "Almost always satisfied (3)" and "Always satisfied (4)". A high score indicates an increase in parental satisfaction.

SECONDARY OUTCOMES:
Physiological Parameter Monitoring Form | Second measurement: 1 minute after treatment
  Heart rate (min), oxygen saturation (SpO2%), blood pressure (mmHg) and respiratory rate (min) were measured one minute after treatment administration.
Children's State Anxiety and Children's Fear Scale | Second measurement: 1 minute after treatment
  1 minute after the treatment, the child's anxiety and fear score was scored again.
Visual Analog Scale | Second measurement: 1 minute after treatment
  One minute after the treatment, the child's pain score was scored again

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Kucukoglu, Prof, Principal Investigator — Selcuk University
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published.

REFERENCES:
- [Background] Bergomi P, Scudeller L, Pintaldi S, Dal Molin A. Efficacy of Non-pharmacological Methods of Pain Management in Children Undergoing Venipuncture in a Pediatric Outpatient Clinic: A Randomized Controlled Trial of Audiovisual Distraction and External Cold and Vibration. J Pediatr Nurs. 2018 Sep-Oct;42:e66-e72. doi: 10.1016/j.pedn.2018.04.011. Epub 2018 May 1. PMID 29728296
- [Background] Silva SGTD, Santos MA, Floriano CMF, Damiao EBC, Campos FV, Rossato LM. Influence of Therapeutic Play on the anxiety of hospitalized school-age children: Clinical trial. Rev Bras Enferm. 2017 Nov-Dec;70(6):1244-1249. doi: 10.1590/0034-7167-2016-0353. English, Portuguese. PMID 29160486
- [Background] Roberts JG, Prys-Roberts C, Foex P, Clarke TN, Bennett M. Proceedings: A comparison of the effects of practolol and propranolol on the response to haemorrhage in anaesthetized dogs after myocardial infarction. Br J Anaesth. 1973 Dec;45(12):1230. doi: 10.1093/bja/45.12.1230. No abstract available. PMID 4787017
- [Background] Kose S, Arikan D. The Effects of Cartoon Assisted Endoscopy Preparation Package on Children's Fear and Anxiety Levels and Parental Satisfaction in Turkey. J Pediatr Nurs. 2020 Jul-Aug;53:e72-e79. doi: 10.1016/j.pedn.2020.02.010. Epub 2020 Mar 13. PMID 32173165
- [Background] Inan G, Inal S. The Impact of 3 Different Distraction Techniques on the Pain and Anxiety Levels of Children During Venipuncture: A Clinical Trial. Clin J Pain. 2019 Feb;35(2):140-147. doi: 10.1097/AJP.0000000000000666. PMID 30362982
- [Background] Masmoudi A, el-Fetouaki J, Weltin D, Belhadj O, Mandel P. Association of mitochondrial ADP-ribosyl transferase activity with the DNA-protein complex. Biochem Mol Biol Int. 1993 Jan;29(1):77-83. PMID 8387848
- [Background] Burns-Nader S, Joe L, Pinion K. Computer tablet distraction reduces pain and anxiety in pediatric burn patients undergoing hydrotherapy: A randomized trial. Burns. 2017 Sep;43(6):1203-1211. doi: 10.1016/j.burns.2017.02.015. Epub 2017 Mar 18. PMID 28318748